CLINICAL TRIAL: NCT06509529
Title: The Effect of Motivational Interviewing Based on the COM-B Model on Women's Cervical Cancer Health Beliefs and Participation in Screening: A Single-Blind Randomized Controlled Study
Brief Title: The Effect of Motivational Interviewing Based on the COM-B Model
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, Hacer Gok Ugur, Associate Professor., Ordu University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Ordu1
Record Dates: First submitted 2024-07-14; First posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Cervical Cancer
Keywords: Cervical Cancer; Motivational Interviewing; Early Diagnosis and Screening; Health Beliefs; Nursing; COM-B Model
MeSH Terms: conditions — Uterine Cervical Neoplasms; Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Motivational interviews based on the COM-B Model will be given to the women in the experimental group.
  Interventions: Other: Motivational Interviewing Based on the COM-B Model
- control group (No Intervention): They will receive routine cancer screening information provided by the institution.

INTERVENTIONS:
Other: Motivational Interviewing Based on the COM-B Model — Motivational Interviewing Based on the COM-B Model will be applied to the women in the experimental group.
  Arms: Experimental group

SUMMARY:
This research will be conducted to determine the effect of motivational interviewing based on the COM-B model on women's cervical cancer health beliefs and participation in screening.

DETAILED DESCRIPTION:
Cancer is an important public health problem in terms of mortality and morbidity in the world and in our country, and ranks second among the causes of death. It can reduce the mortality and morbidity rate in cancer with early diagnosis and screening studies. One of the cancers for which early diagnosis and screening studies are carried out in women is cervical cancer, and it is the 4th most frequently diagnosed cancer type that causes death in women. Although early diagnosis and screening studies are carried out, women do not participate in enough cervical cancer screenings for different reasons. Interventions are needed to increase women's motivation to participate in screening. This research will be conducted to determine the effect of motivational interviewing based on the COM-B model on women's cervical cancer health beliefs and participation in screening. The research is planned as a parallel group single-blind randomized controlled experimental study and will be conducted on women between the ages of 30-65 who are registered at Altınordu Central Family Health Center in Ordu Province. The population of the research will be women between the ages of 30-65 who are registered at Altınordu Central Family Health Center, and the sample will be 74 women who meet the research criteria and agree to participate in the research. The data of the research will be collected with the "Information Form", "Cervical Cancer and Pap Smear Test Health Belief Model Scale", "Cervical Cancer Screening Status Evaluation Form" and "Satisfaction Evaluation Form". A motivational interview program based on the COM-B Model will be applied to the women in the experimental group for 1 month (1st week face-to-face, 2nd, 3rd and 4th weeks online). No intervention will be applied to the control group during the research process. The analysis of the data will be done in a computer environment by an expert statistician. Necessary institutional permissions and ethics committee approval will be obtained for the research.

ELIGIBILITY:
Inclusion Criteria:

* Registered at Altınordu Central Family Health Center,
* A woman,
* Between 30-65 years of age,
* The one who is married,
* Have not had a Pap Smear test in the last 5 years,
* Has a smart phone
* Has an internet connection,
* Open to communication and collaboration,
* Women who volunteer to participate in the study will be included in the study.

Exclusion Criteria:

* Who had total hysterectomy surgery,
* The pregnant one,
* Those diagnosed with cervical cancer and
* Women with a psychiatric diagnosis will be excluded from the study.

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 68 (Estimated)
Dates: Start 2024-08-15 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
"Cervical Cancer and Pap Smear Test Health Belief Model Scale" | 0th month and 1st month.
  The scale was developed by Güvenç et al. (2011). Higher scores from the scale indicate increased sensitivity, caring and motivation; It indicates that benefits are perceived as high for benefit perception and obstacles are perceived as high for obstacle perception.
Status of Cervical Cancer Screening | 0th month and 1st month.
  This form was prepared by the researcher and will evaluate women's status of being screened for cervical cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Hacer GÖK UĞUR, Assoc.Prof., Study Director — Ordu University

IPD SHARING:
Plan to Share IPD: No